CLINICAL TRIAL: NCT05310513
Title: The Predictors of ICU Admission of Obstetric Posterion Reversible Encephalopathy Syndrome
Brief Title: The Predictors of ICU Admission of oPRES
Status: Completed | Type: Observational
Sponsor: Dunjin Chen (Other)
Responsible Party: Sponsor-Investigator, Dunjin Chen, Director of obstetrics, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Other Study IDs: 2019A151510102
Record Dates: First submitted 2022-03-15; First posted 2022-04-05 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Posterior Reversible Encephalopathy Syndrome; Intensive Care Units
MeSH Terms: conditions — Posterior Leukoencephalopathy Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU group: patients admitted to ICU with PRES.
  Interventions: Other: Whether the patient needs to be admitted to the ICU
- Non-ICU group: patients not admitted to ICU with PRES.
  Interventions: Other: Whether the patient needs to be admitted to the ICU

INTERVENTIONS:
Other: Whether the patient needs to be admitted to the ICU — According to ICU admission or not, patients were grouped into ICU group and NOT-ICU group.

SUMMARY:
The purpose of this study is to explore the predictors of ICU admission of obstetric posterior reversible encephalopathy syndrome.

DETAILED DESCRIPTION:
The investigators retrospectively collected data (General information, clinical data, biochemical indicators, imaging features, and pregnancy outcome) from pregnant woman diagnosed with PRES to explore the predictors of ICU admission during 2012 to 2021.Then, the investigators grouped all the patients into ICU group and Non-ICU group according to ICU admission or not.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant Women were diagnosed of PRES.
2. all patients provided written informed consent

Exclusion Criteria:

1. patients combined with other neurological disorders
2. patients combined with mental illness

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant Women diagnosed with PRES
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure(BP) | The BP of patients was obtained immediately at the onset of symptoms.
  blood pressure including systolic blood pressure (SBP), and diastolic blood pressure (DBP).
severity of the edema | Cranial Imaging was examined immediately at the onset of symptoms, such as s headaches, visual changes, seizures, consciousness impairment.
  The extent and severity of the edema observed in the lesion area were graded on a scale of 0-5 by evaluating FLAIR images.(0, normal; 1, limited cortical or subcortical white matter oedema; 2, white matter oedema > cortical oedema, white matter oedema extending into deep white matter; 3, white matter oedema > cortex oedema, oedema extending to the ventricular surface; 4, the involved regions substantially extend to the ventricular surface and are almost com- pletely conﬂuent; 5, involved regions are fully conﬂuent and con- tinuous, ventricular deformity due to the oedema).
pregnancy outcomes | The pregnancy outcomes will record immediately when the patients deliver.
  The rates of stillbirth and premature birth (gestation less than 37 weeks) in PRES patients.
biochemical parameters | Biochemical indicators were collected within 1 week of the hospital stay.
  The level of lactate dehydrogenase(LDH) will be measured，and LDH﹥380U/L means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dunjin Chen, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Obstetrics and Gynecology, Key Laboratory for Major Obstetric Diseases of Guangdong Province, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No